CLINICAL TRIAL: NCT06999681
Title: A Prospective Study on the Association of Perioperative Echocardiographic Parameters and Other Risk Factors With Postoperative Atrial Fibrillation
Brief Title: Postoperative Arrhythmia and Preoperative Cardiac Function
Status: Not yet recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, National Taiwan University Clinical Trial Center, Attending anesthesiologist, National Taiwan University Hospital
Other Study IDs: 202505037RINE
Record Dates: First submitted 2025-05-22; First posted 2025-05-31 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: The Cardiac Function
Keywords: cardiac echo; cardiac surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with postoperative arrhythmia: patients with postoperative arrhythmia after cardiac surgery
  Interventions: Other: No Interventions
- patients without postoperative arrhythmia: patients without postoperative arrhythmia after cardiac surgery
  Interventions: Other: No interventions

INTERVENTIONS:
Other: No Interventions — this is an observational cohort study. There was no intervention.
  Groups: patients with postoperative arrhythmia
Other: No interventions — No interventions in this study. This study is an observational study.
  Groups: patients without postoperative arrhythmia

SUMMARY:
This study aims to investigate the association between echocardiographic parameters-including preoperative cardiac echo, as well as postoperative follow-up echocardiography and other associated parameters-and the risk factors related to postoperative arrhythmia

DETAILED DESCRIPTION:
Postoperative atrial fibrillation (POAF), defined as newly onset atrial fibrillation occurring during hospitalization, is a common complication following cardiac surgery, affecting approximately 20-30% of patients. Studies have shown that patients who develop POAF experience longer hospital stays, incur higher medical costs, and have increased rates of stroke- and heart failure-related complications, as well as higher risks of readmission and mortality.

POAF is generally believed to result from acute perioperative triggers acting on preexisting structural abnormalities of the atria or ventricles. However, the echocardiographic predictors of POAF remain poorly understood. While previous studies have examined the association between preoperative transthoracic echocardiography (TTE)-assessed left atrial and left ventricular function and the development of POAF, the detailed relationship between intraoperative transesophageal echocardiography (TEE)-assessed atrial and ventricular function, its intraoperative changes, and POAF remains insufficiently explored.

This study aims to investigate the association between echocardiographic parameters-including preoperative TTE and TEE, as well as postoperative follow-up parameters-and the risk factors related to POAF.

ELIGIBILITY:
Inclusion Criteria:

* patients receiving cardiac surgery

Exclusion Criteria:

* preoperative arrhythmia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing cardiac surgery
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-05-26 (Estimated); Primary Completion 2030-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
The occurrence of postoperative arrhythmia | postoperative 1 years
  postoperative arrhythmia after cardiac surgery

IPD SHARING:
Plan to Share IPD: No
Due to ethical issue